CLINICAL TRIAL: NCT04092088
Title: Effectiveness of Cerebral and Peripheral Electrical Stimulation on Pain and Functional Limitations Associated With Carpal Tunnel Syndrome: A Randomized, Double-blind, Multi-center, Factorial Clinical Trial
Brief Title: Effects of Cerebral & Peripheral Electrical Stimulation on Pain and Function in CTS
Acronym: DCS-ENS-CTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suez Canal University (Other)
Collaborators: Hiroshima University (Other); Complejo Hospitalario de Especialidades Juan Ramón Jimenez (Other); Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim El-Sayed Maaty, Principal investigator, Suez Canal University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: AIMAATY
Record Dates: First submitted 2019-07-13; First posted 2019-09-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Transcranial Direct Current Stimulation (tDCS); Transcutaneous Electrical Nerve Stimulation (TENS); analgesic effect; functional disability
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Transcranial Direct Current Stimulation; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: randomized, triple-blind, multi-center, factorial clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: neither the participant nor the investigator and outcomes assessor will be aware whether active tDCS/TENS will be applied to a particular case.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- tDCS-r+TENS-r (Active Comparator): Real transcranial direct current stimulation (tDCS-r) + real transcutaneous electrical nerve stimulation (TENS-r)
  Interventions: Device: tDCS-r; Device: TENS-r
- tDCS-r+TENS-s (Experimental): Real transcranial direct current stimulation (tDCS-r) + sham transcutaneous electrical nerve stimulation (TENS-s)
  Interventions: Device: tDCS-r; Device: TENS-s
- tDCS-s+TENS-r (Experimental): Sham transcranial direct current stimulation (tDCS-s) + real transcutaneous electrical nerve stimulation (TENS-r)
  Interventions: Device: TENS-r; Device: tDCS-s
- tDCS-s+TENS-s (Sham Comparator): Sham transcranial direct current stimulation (tDCS-s) + sham transcutaneous electrical nerve stimulation (TENS-s)
  Interventions: Device: tDCS-s; Device: TENS-s

INTERVENTIONS:
Device: tDCS-r — The transcranial stimulation will be applied by a constant current device (tdcs) with an intensity of 2 mA for 20 minutes (the set will be turned on for 20 minutes).
  Other Names: real (active) transcranial direct current stimulation
  Arms: tDCS-r+TENS-r; tDCS-r+TENS-s
Device: TENS-r — Conventional TENS will be applied for 20 minutes. The cathode will be placed on the carpal ligament, and the anode electrodes on the palmar area of the hand, with a layer of conductive gel applied to the area (the set will be turned on for 20 minutes)..
  Other Names: real (active) transcutaneous electrical nerve stimulation
  Arms: tDCS-r+TENS-r; tDCS-s+TENS-r
Device: tDCS-s — The transcranial stimulation will be applied by a constant current device (tdcs) with an intensity of 2 mA for 20 minutes (the set will be turned off after 30 seconds).
  Other Names: sham transcranial direct current stimulation
  Arms: tDCS-s+TENS-r; tDCS-s+TENS-s
Device: TENS-s — Conventional TENS will be applied for 20 minutes. The cathode will be placed on the carpal ligament, and the anode electrodes on the palmar area of the hand, with a layer of conductive gel applied to the area (the set will be turned off after 30 seconds).
  Other Names: sham transcutaneous electrical nerve stimulation
  Arms: tDCS-r+TENS-s; tDCS-s+TENS-s

SUMMARY:
This is a randomized, double-blind, multi-center, factorial clinical trial to study the effectiveness of cerebral and peripheral electrical stimulation on pain and functional limitations associated with carpal tunnel syndrome (CTS). The study subjects will be randomly into four groups; (1) active trans-cranial direct current stimulation (tDCS) + active trans-cutaneous electrical nerve stimulation (TENS), (2) active tDCS + sham TENS, (3) sham tDCS + active TENS and (4) sham tDCS + sham TENS. The patient will be assessed by Brief Pain Inventory (BPI), Beck Depression Inventory (BDI), The Douleur Neuropathique en 4 questions (DN4), Quantitative sensory testing (QST), Pain Pressure Test (PPT) with algometer, Conditioned pain modulation (CPM), Patient ratings of improvement, or worsening, of the pain condition, Quality of Life short-form (SF)-36, Visual Analog Mood Scale (VAMS), Mini Mental Status Exam (MMSE) and Adverse Events Questionnaire (AEs). This study aims to investigate whether cerebral and peripheral electrical stimulation combined are more effective in relieving pain and functional limitations than the separate application of electrical stimulation in patients with CTS.

DETAILED DESCRIPTION:
The study will be carried out on patients attending (1) Physical Medicine, Rheumatology and Rehabilitation outpatient clinic in Suez Canal University Hospital, Ismailia, EGYPT, (2) Hiroshima University, (3) Department of Physical Medicine & Rehabilitation, Juan Ramón Jiménez University Hospital, Huelva, Spain, and (4) University of Sherbrooke, Canada and diagnosed with CTS according to clinical examination and to the American Association of Neuromuscular and Electrodiagnostic Medicine (AANEM) practice recommendations for CTS.

Study subjects will be divided into four groups:

Group (1): (active comparator = tDCS-real (r) + TENS-r) will include 45 patients with CTS and will receive active anodal tDCS of M1 for 20 minutes, at 2 mA plus active TENS (the cathode will be placed on the carpal ligament, and the anode electrodes on the palmar area of the hand) for 20 minutes, and a total of 15 sessions for 3 weeks (5 per week) will be completed.

Group (2): (experimental group= tDCS-r + TENS-sham (s)) will include 45 patients with CTS and will receive active tDCS M1 for 20 minutes plus sham TENS for 20 minutes, and a total of 15 sessions for 3 weeks (5 per week).

Group (3): (experimental group= tDCS-s + TENS-r) will include 45 patients with CTS and will receive sham tDCS M1 for 20 minutes (the set will be turned off after 30 seconds) plus active TENS for 20 minutes, and a total of 15 sessions for 3 weeks (5 per week).

Group (4): (sham comparator = tDCS-s + TENS-s) will include 45 patients with CTS and will receive sham tDCS M1 for 20 minutes (the set will be turned off after 30 seconds) plus sham TENS for 20 minutes, and a total of 15 sessions for 3 weeks (5 per week).

The study sample will be collected from all patients with CTS fulfilling the eligibility criteria, will be eligible to join the study (either referred for electrophysiological study or presented to the clinic for primary assessment). To make sure that no bias should enter the assessment of the results, neither the patient nor the clinicians will be aware whether active tDCS/TENS will be applied to a particular case. To ensure this result, one symbol of these four symbols (square, circle, star and triangle) will be applied to one group of the four groups in the physiotherapy sheet and only the physiotherapist knew the key for each symbol. At the end of the study, the four groups will be revealed in order to analyze the results according to proper statistical measures.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged >18 years and <65 years.
* Paresthesia, pain or vasomotor symptoms through the distribution of median nerve (persistence > 2 months).
* Positive result for Phalen's, Tinel's and/or carpal compression tests during physical examination.
* Mild-to-moderate severity of CTS according to American Association of Neuromuscular & Electrodiagnostic Medicine (AANEM) 2002 (mild: abnormal sensory peak latency [≥3.5ms] with normal motor distal latency [<4.4]; moderate: abnormal sensory [≥3.5ms] and motor [≥4.4ms] latencies).

Exclusion Criteria:

* Previous history of wrist surgery
* Presence of predisposing etiological factors for CTS (e.g., diabetes mellitus).
* Trauma, neurological, psychiatric, rheumatic diseases, renal failure, pregnancy, hypothyroidism, and hyperthyroidism.
* Presence of conditions that might cause numbness in the hand, including cervical radiculopathy, cervical ribs, plexopathy, and polyneuropathy.
* Pharmacological treatment with oral steroids or non-steroidal anti-inflammatory drugs within the previous month.
* Participation in a physical therapy program.
* Administration of steroid injection(s) within the previous 6 months.
* Previous treatment with TENS <6 months.
* Previous treatment with tDCS.
* Use of pacemakers or other implanted devices.
* Pregnancy or breastfeeding.
* Refuse to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | At baseline
  A short, self-report questionnaire includes 4 items that assess pain intensity (pain right now, pain on average in last 24 hours, worst pain in last 24 hours, and least pain in last 24 hours) using an NRS from 0 (no pain) to 10 (pain as bad as can imagine). The mean of these 4 pain items will be used as primary outcome. The BPI also includes 7 items that assess the impact of the pain on functioning using a 0 (no interference) to 10 (complete interference) rating scale, which will be used as a secondary outcome.
Brief Pain Inventory (BPI) | After 3 weeks
  A short, self-report questionnaire includes 4 items that assess pain intensity (pain right now, pain on average in last 24 hours, worst pain in last 24 hours, and least pain in last 24 hours) using an NRS from 0 (no pain) to 10 (pain as bad as can imagine). The mean of these 4 pain items will be used as primary outcome. The BPI also includes 7 items that assess the impact of the pain on functioning using a 0 (no interference) to 10 (complete interference) rating scale, which will be used as a secondary outcome.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | At baseline
  To assess depressive symptoms by using the 21-item The cut-off point for depression is set at 9/10 (normal mood, scores 0-9 vs. elevated depressions symptoms, scores 10 or more).
Beck Depression Inventory (BDI) | After 3 weeks
  To assess depressive symptoms by using the 21-item The cut-off point for depression is set at 9/10 (normal mood, scores 0-9 vs. elevated depressions symptoms, scores 10 or more).
The Douleur Neuropathique 4 questions (DN4) | At baseline
  A simple and objective tool, primarily designed to screen for neuropathic pain, differentiating between neuropathic and nociceptive pain conditions in clinical practice and research studies. In total, it contains 10 questions with a binary answer (no/yes). The total score, ranging from 0 to 10, is obtained by adding the number of affirmative answers, a total score > 4 out of 10 suggests neuropathic pain.
The Douleur Neuropathique 4 questions (DN4) | After 3 weeks
  A simple and objective tool, primarily designed to screen for neuropathic pain, differentiating between neuropathic and nociceptive pain conditions in clinical practice and research studies. In total, it contains 10 questions with a binary answer (no/yes). The total score, ranging from 0 to 10, is obtained by adding the number of affirmative answers, a total score > 4 out of 10 suggests neuropathic pain.
Quantitative sensory testing (QST) | At baseline
  The Semmes-Weinstein Monofilament test kit will be used to evaluate sensory thresholds of the tips of the thumb, the index, and the middle fingers. The kit consists of 20 flexible nylon monofilaments of varying diameter and length to measure the level of skin touch sensation. The monofilaments have log numbers from 1.65 to 6.65 which begins with the light filaments (1.65-3.61) and progresses to heavy filaments of increasing diameter (3.84-6.65). Heavy filaments need increased pressure for touch to be recognized by patients. The tester applies each monofilament to the surface area of the skin with a perpendicular angle, then applies slight and steady pressure until the monofilament begins to bend, which is the end point of the test. The monofilament number 2.83 was defined as cut-off for normal sensation.
Quantitative sensory testing (QST) | After 3 weeks
  The Semmes-Weinstein Monofilament test kit will be used to evaluate sensory thresholds of the tips of the thumb, the index, and the middle fingers. The kit consists of 20 flexible nylon monofilaments of varying diameter and length to measure the level of skin touch sensation. The monofilaments have log numbers from 1.65 to 6.65 which begins with the light filaments (1.65-3.61) and progresses to heavy filaments of increasing diameter (3.84-6.65). Heavy filaments need increased pressure for touch to be recognized by patients. The tester applies each monofilament to the surface area of the skin with a perpendicular angle, then applies slight and steady pressure until the monofilament begins to bend, which is the end point of the test. The monofilament number 2.83 was defined as cut-off for normal sensation.
Pain Pressure Test (PPT) with algometer | At baseline
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure where a sense of pressure first changes to pain. An electronic algometer will be used to measure PPT levels. The algometer consists of a 1 cm2 rubber-tipped plunger mounted on a force transducer. The pressure is applied approximately at a rate of 30 kPa/s, with the algometer placed perpendicular to the application point. Participants will be instructed to press switch when the sensation changed from pressure to pain. The mean of three trials (intra-examiner reliability) will be calculated and used for main analysis. A 30 s resting period will be allowed between each measure.
Pain Pressure Test (PPT) with algometer | After 3 weeks
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure where a sense of pressure first changes to pain. An electronic algometer will be used to measure PPT levels. The algometer consists of a 1 cm2 rubber-tipped plunger mounted on a force transducer. The pressure is applied approximately at a rate of 30 kPa/s, with the algometer placed perpendicular to the application point. Participants will be instructed to press switch when the sensation changed from pressure to pain. The mean of three trials (intra-examiner reliability) will be calculated and used for main analysis. A 30 s resting period will be allowed between each measure.
Conditioned pain modulation (CPM) | At baseline
  A CPM paradigm with the cold pressor test will be was used. Participants will submerge one foot into an insulated container filled with cold water with the medial malleolus ~3 cm below the water line. The foot contralateral to the affected hand (or most affected hand in case of bilateral CTS) will be submerged. Participants will rate the cold-induced foot pain on a numric pain rating scale (NPRS), ranging from 0 (no pain) to 10 (worst pain imaginable). Immediately after maintaining the NPRS within the target score for 30 seconds, the test stimulus will be given. Pressure pain threshold (PPT) testing will be applied as a test stimulus. PPTs will be measured with a digital algometer. The participants will press a button as soon as the sensation of pressure changed to pain. PPT measurements will be taken on the thenar and hypothenar eminence of both hands, before cold water immersion and during cold water immersion.
Conditioned pain modulation (CPM) | After 3 weeks
  A CPM paradigm with the cold pressor test will be was used. Participants will submerge one foot into an insulated container filled with cold water with the medial malleolus ~3 cm below the water line. The foot contralateral to the affected hand (or most affected hand in case of bilateral CTS) will be submerged. Participants will rate the cold-induced foot pain on a numric pain rating scale (NPRS), ranging from 0 (no pain) to 10 (worst pain imaginable). Immediately after maintaining the NPRS within the target score for 30 seconds, the test stimulus will be given. Pressure pain threshold (PPT) testing will be applied as a test stimulus. PPTs will be measured with a digital algometer. The participants will press a button as soon as the sensation of pressure changed to pain. PPT measurements will be taken on the thenar and hypothenar eminence of both hands, before cold water immersion and during cold water immersion.
Patient ratings of improvement, or worsening, of the pain condition | At baseline
  Patient's Clinical Global Impression of Change scale, subjects select one of seven options describing response to treatment, ranging from 1-7 where 1 indicates "very much improved" and 7 indicates "very much worse.".
Patient ratings of improvement, or worsening, of the pain condition | After 3 weeks
  Patient's Clinical Global Impression of Change scale, subjects select one of seven options describing response to treatment, ranging from 1-7 where 1 indicates "very much improved" and 7 indicates "very much worse.".
Quality of Life short-form-36 | At baseline
  To assess quality of Life, it consists of 36 items divided into eight domains range from reflecting predominantly physical well-being, that include physical function, the ability to perform expected physical roles, the degree of bodily pain and overall sense of general health to those reflecting predominantly social and emotional well-being that include overall sense of vitality, ability to function in social roles, ability to perform expected emotional and social roles and overall sense of mental health. Each item has 5 response choices, a high score (response choice 5) and a low score (response choice 1).
Quality of Life short-form-36 | After 3 weeks
  To assess quality of Life, it consists of 36 items divided into eight domains range from reflecting predominantly physical well-being, that include physical function, the ability to perform expected physical roles, the degree of bodily pain and overall sense of general health to those reflecting predominantly social and emotional well-being that include overall sense of vitality, ability to function in social roles, ability to perform expected emotional and social roles and overall sense of mental health. Each item has 5 response choices, a high score (response choice 5) and a low score (response choice 1).
Visual Analog Mood Scale | At baseline
  A self-assessment scale in which subjects rate their own emotions, including anxiety, depression, stress, and sleepiness along a 100 mm line.
Visual Analog Mood Scale | After 3 weeks
  A self-assessment scale in which subjects rate their own emotions, including anxiety, depression, stress, and sleepiness along a 100 mm line.
Mini Mental Status Exam | At baseline
  Cognition will be analyzed using Mini-Mental Status Examination, a brief screening of cognitive abilities.
Mini Mental Status Exam | After 3 weeks
  Cognition will be analyzed using Mini-Mental Status Examination, a brief screening of cognitive abilities.
Adverse Events Questionnaire | After 3 weeks
  At each stimulation session and all follow-ups, participants will be administered a questionnaire to evaluate the potential adverse effects of stimulation on a 5-point scale from 0-4 (0 indicates no adverse events and 4 indicates extreme adverse effects. The main potential adverse effects include headache, neck and scalp pain, tingling, sleepiness, and acute mood change.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed I Maaty, MD, Principal Investigator — Suez Canal University

IPD SHARING:
Plan to Share IPD: Yes
Informed consent, data management and statistical analysis will shared, if requested, through the investigator e-mail.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available after the end of the study
Access Criteria: Informed consent, data management and statistical analysis will shared, if requested, through e-mail: aimaaty@hotmail.com